CLINICAL TRIAL: NCT07400276
Title: Ayurveda-inspired Diet and Lifestyle Intervention for Glycemic, Anthropometric, and Stress Improvements in Type 2 Diabetes: A Feasibility Study
Brief Title: Ayurveda Diet & Lifestyle Protocol for Type 2 Diabetes: A Feasibility Study
Acronym: AYU-LIFE-T2D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi International University (Other)
Responsible Party: Principal Investigator, Amandeep Negi, Doctoral Researcher, Maharishi International University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Approval 2025_02_8
Record Dates: First submitted 2026-02-02; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Ayurveda; Type 2 Diabetes Mellitus; Diet & Lifestyle Intervention; Maharishi Yoga Asanas; Bhramari Pranayama; Feasibility Study
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This was a single-group feasibility study evaluating the acceptability, adherence, and implementation of a multi-component lifestyle intervention delivered alongside usual medical care. The study was not designed to test comparative efficacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ayurveda Lifestyle Program (Experimental): Participants in this single-arm feasibility study received a 12-week Maharishi Ayurveda-based lifestyle program that integrated dietary and lifestyle guidance, yoga-based physical activity, and breathing practices. All participants assigned to this arm received the same intervention and were followed for feasibility, adherence, and health-related outcomes.
  Interventions: Behavioral: Maharishi Ayurveda Lifestyle Program

INTERVENTIONS:
Behavioral: Maharishi Ayurveda Lifestyle Program — A 12-week integrative behavioral lifestyle program combining
  1. an Ayurvedic Diabetic Diet and Reset (DDR) Plan emphasizing low-glycemic-index food choices, meal regularity, and health-related lifestyle behaviors aligned with Ayurvedic principles;
  2. guided Maharishi Yoga Asanas; and
  3. daily Bhramari Pranayama breathing practice. The program was supported through scheduled phone and text check-ins.
  Other Names: Ayurvedic Diabetic Diet and Reset (DDR) Plan; Maharishi Yoga Asanas; Bhramari Pranayama

SUMMARY:
This study looked at whether a 12-week Maharishi Ayurveda diet and lifestyle program was practical and acceptable for adults with Type 2 Diabetes. The program was offered through Family Health Centers in North Carolina and combined three parts: an Ayurvedic-based diet plan, guided yoga postures, and a breathing practice.

Seventeen participants started the program, and twelve completed the full 12- week intervention. The study focused on whether participants were able to follow the program regularly, complete study activities, and stay in the study for the full period. Participants were asked to practice the program at least five days per week and received regular support through scheduled and as-needed communication via phone, text messages, email, and video-based materials throughout the study.

The study also tracked changes in daily health habits, blood sugar levels, body weight, waist size, stress, and diabetes-related emotional well-being. Some information was collected using questionnaires, and some measurements were taken through clinic visits or home glucose monitoring.

Most participants who completed the program were able to follow the activities as instructed. Changes were observed in blood sugar levels, body weight, waist size, and measures of stress and diabetes-related distress. No serious safety concerns were reported.

Overall, the study showed that this Ayurvedic diet and lifestyle program could be safely carried out in a primary care setting. The results support further research with larger groups to better understand its potential benefits over time.

DETAILED DESCRIPTION:
Background and Rationale:

Type 2 Diabetes Mellitus (T2DM) is a chronic condition influenced by both genetic and modifiable lifestyle factors, including diet, physical inactivity, stress, and obesity. In the United States, diabetes prevalence has increased substantially over the past two decades, in part due to lifestyle-related factors. Although pharmacological therapies are widely used, long-term diabetes management remains challenging because of adherence difficulties, side effects, and psychosocial burden. Integrative lifestyle approaches that incorporate dietary regulation, physical activity, and stress-reduction practices may support diabetes self-management; however, their feasibility and acceptability within U.S. primary care settings require further evaluation.

Study Objective The primary objective of this study was to assess the feasibility, acceptability, and safety of a 12-week Maharishi Ayurveda-inspired diet and lifestyle program for adults with T2DM. The study aimed to evaluate participant adherence, program completion, and the practicality of implementing this multi-component intervention in a real-world primary care context.

Study Design This was a single-arm feasibility study conducted at Family Health Centers in North Carolina, USA. Adults with a diagnosis of T2DM were recruited from the clinic population. Seventeen participants initiated the intervention, and twelve completed the full 12-week program.

Intervention Overview

Participants received a structured 12-week lifestyle intervention consisting of three integrated components:

Dietary Component The Ayurvedic Diabetic Diet and Reset (DDR) Plan emphasized low-glycemic-index food choices, meal regularity, and dietary patterns aligned with Ayurvedic principles of digestive balance and broader health-related lifestyle behaviors. The plan focused on food categories, preparation methods, and meal timing rather than caloric prescription. During the dietary reset phase (approximately Weeks 1-8), participants were progressively introduced to core DDR principles, food lists, and simplified recipes to support gradual dietary transition and feasibility. Study-specific recipes and educational materials were delivered through recorded video modules.

Physical Activity Component Maharishi Yoga Asanas (MYA) consisted of a standardized sequence of physical postures designed to support physical mobility, circulation, and stress regulation. Participants were trained using video-based instruction and received remote guidance as needed throughout the intervention period.

Breathing Practice Bhramari Pranayama, a slow humming breath practice, was included to support stress regulation. Participants were instructed to practice daily following Maharishi Yoga Asanas, beginning with approximately five minutes per session and progressing to ten minutes over the course of the intervention.

Adherence Monitoring and Support Participants were instructed to engage in the intervention components at least five days per week. Daily engagement was self-monitored using SMART (Self-Monitoring and Review Tracking) log sheets, which were completed daily and submitted to the study team every two weeks. Adherence support and clarification were provided through scheduled text messages and phone calls approximately every one to two weeks, with additional communication as needed. Intervention materials were delivered digitally. Participants used home glucometers to self-monitor fasting blood glucose, with readings reported biweekly during the intervention period.

ELIGIBILITY:
Inclusion Criteria

* Adults aged 18 to 70 years
* Diagnosed with Type 2 Diabetes Mellitus
* Hemoglobin A1c between 6.5% and 9.5%
* Receiving primary care at the Family Health Centers in North Carolina
* Stable oral diabetes medication regimen for at least 3 months prior to enrollment
* Able and willing to follow the study diet, yoga, and breathing practices
* Able to communicate in English
* Able to provide informed consent

Exclusion Criteria

* Diagnosis of Type 1 Diabetes
* Current use of insulin
* Recent changes in diabetes medications within the past 3 months
* Pregnant or breastfeeding
* Uncontrolled psychiatric illness that would interfere with participation
* Physical limitations that prevent participation in yoga or movement practices
* History of eating disorders
* Allergy or strong aversion to foods used in the study diet
* Participation in another lifestyle or intervention study during the study period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2025-05-02 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
Change in Health Habits Assessment Scale (HHAS) Score | Baseline, 6 weeks, and 12 weeks
  The HHAS is a self-report measure developed to assess participant engagement in health-promoting habits, including dietary choices, physical activity, daily routine, and stress-reduction practices. In this study, it was used to evaluate the feasibility and behavioral adherence to the Maharishi Ayurveda-based lifestyle program. Participants completed the HHAS at baseline, mid-, and post-intervention.

SECONDARY OUTCOMES:
Change in Hemoglobin A1c (HbA1c) | Baseline and 12 weeks
  HbA1c was measured in a CLIA-certified lab at the Family Health Centers at baseline and after 12 weeks to assess longer-term glycemic control. This was a key clinical biomarker for evaluating the physiological impact of the diet & lifestyle intervention.
Change in Fasting Blood Glucose (FBG) | Baseline, 2, 4, 6, 8, 10, and 12 weeks
  FBG was assessed through CLIA-certified laboratory tests at baseline and at 12 weeks. Additionally, participants used home glucometers to measure FBG at 2, 4, 6, 8, 10, and 12 weeks. These combined measures were used to evaluate short-term glycemic response to the lifestyle intervention.
Change in Body Weight (in lbs.) | Baseline and 12 weeks
  Body weight was measured in pounds (lbs.) and converted to kilograms (kg) for analysis. Measurements were taken using standard calibrated clinical scales at the Family Health Centers.
Change in Body Waist Circumference (WC) | Baseline and 12 weeks
  Waist circumference was measured (in inches) at baseline and 12 weeks to assess changes in anthropometric indicators associated with metabolic health. Measurements were taken using standard clinical tools at the Family Health Centers.
Change in Body Mass Index (BMI) | Baseline and 12 weeks
  Body Mass Index (BMI) was calculated using height and weight measurements obtained by Family Health Centers' clinical staff at baseline and post-intervention. BMI values were expressed in kilograms per square meter (kg/m²).

OTHER OUTCOMES:
Change in Perceived Stress Scale-10 (PSS-10) Score | Baseline, 6 weeks, and 12 weeks
  The Perceived Stress Scale-10 (PSS-10) is a validated questionnaire used to measure perceived stress levels over the past month. Participants completed the scale at baseline, 6 weeks, and 12 weeks to evaluate psychological changes during the 12-week Ayurvedic lifestyle intervention.
Change in Problem Areas in Diabetes (PAID) Score | Baseline, 6 weeks, and 12 weeks
  The Problem Areas in Diabetes (PAID) scale is a validated tool assessing emotional distress related to diabetes management. Participants completed the PAID scale at baseline, 6 weeks, and 12 weeks to measure changes in diabetes-related emotional burden over the course of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Amandeep Negi, BAMS, MHA, Principal Investigator — Maharishi International University
Locations (1):
- Family Health Centers, Asheville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
The study team intends to publish results in peer-reviewed journals. A final decision about sharing individual participant data (IPD) has not yet been made. Any future sharing will depend on participant consent, IRB approval, and institutional policies.

REFERENCES:
- [Background] Barclay AW, Petocz P, McMillan-Price J, Flood VM, Prvan T, Mitchell P, Brand-Miller JC. Glycemic index, glycemic load, and chronic disease risk--a meta-analysis of observational studies. Am J Clin Nutr. 2008 Mar;87(3):627-37. doi: 10.1093/ajcn/87.3.627. PMID 18326601
- [Background] Koenigsberg MR, Corliss J. Diabetes Self-Management: Facilitating Lifestyle Change. Am Fam Physician. 2017 Sep 15;96(6):362-370. PMID 28925635
- [Background] Marcy TR, Britton ML, Harrison D. Identification of barriers to appropriate dietary behavior in low-income patients with type 2 diabetes mellitus. Diabetes Ther. 2011 Mar;2(1):9-19. doi: 10.1007/s13300-010-0012-6. Epub 2011 Jan 21. PMID 22127765